CLINICAL TRIAL: NCT02465437
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Multicenter Study to Evaluate Safety, Tolerability, Efficacy, and Pharmacokinetics of JBT-101 in Diffuse Cutaneous Systemic Sclerosis
Brief Title: Safety, Tolerability, Efficacy, and Pharmacokinetics of JBT-101 in Systemic Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated open-label extension
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JBT101-SSc-001
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: JBT-101, Lenabasum, Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- JBT-101 5 mg/20 mg bid (Experimental): JBT-101 5 mg q am and placebo q pm on Days 1-28, then JBT-101 20 mg twice a day (bid) on Days 29-84.
  Interventions: Drug: JBT-101; Drug: Placebo
- JBT-101 20 mg/20 mg bid (Experimental): JBT-101 20 mg q am and placebo q pm on Days 1-28, then JBT-101 20 mg bid on Days 29-84.
  Interventions: Drug: JBT-101; Drug: Placebo
- JBT-101 20 mg bid/20 mg bid (Experimental): JBT-101 20 mg bid on Days 1-84.
  Interventions: Drug: JBT-101
- Placebo (Placebo Comparator): Placebo bid on Days 1-84.
  Interventions: Drug: Placebo
- Part B Open-label (Experimental): JBT-101 20 mg bid on Days 1-364
  Interventions: Drug: Part B Open-Label Extension

INTERVENTIONS:
Drug: JBT-101 — JBT-101 5 mg q am, 20 mg q am, or 20 mg bid on Days 1-28. JBT-101 20 mg bid on Days 29-84.
  Arms: JBT-101 20 mg bid/20 mg bid; JBT-101 20 mg/20 mg bid; JBT-101 5 mg/20 mg bid
Drug: Placebo — Placebo q pm (with JBT-101 5 or 20 mg q AM) or placebo bid on Days 1-28. Placebo bid on Days 29-84.
  Arms: JBT-101 20 mg/20 mg bid; JBT-101 5 mg/20 mg bid; Placebo
Drug: Part B Open-Label Extension — JBT-101 20mg bid on Days 1-364
  Arms: Part B Open-label

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and efficacy of JBT-101 in adult subjects with diffuse cutaneous systemic sclerosis.

DETAILED DESCRIPTION:
Part A of the study is an interventional, double-blind, randomized, placebo-control design will be used to test safety, tolerability, pharmacokinetics, and efficacy of JBT-101 in subjects ≥ 18 and ≤ 70 years of age with active diffuse cutaneous systemic sclerosis. The screening period is up to 28 days, with 84 days treatment period and 28 days follow-up off active treatment.

Part B of the study is an interventional, open-label design will be used. All subjects who complete dosing in Part A without permanent discontinuation of study drug and who pass repeat safety screening will be eligible for enrollment. The screening period is up to 28 days, with a 364 day treatment period and 28 day follow up after last dose of JBT-101.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Diffuse cutaneous systemic sclerosis
* Have skin thickening from SSc in a body area suitable for repeat biopsy
* Disease duration ≤ 3 years from the first non-Raynaud's phenomenon or >3 years and ≤ 6 years from the first non-Raynaud's phenomenon and high sensitivity C-reactive protein > 3 mg/L, high sensitivity interleukin-6 > 5 pg/mL, or increase in mRSS ≥ 5 points over the last 6 months with total RSS ≥ 12.
* Stable treatment for SSc for at least 28 days before Visit 1

Part B

•Completion of dosing in Part A without permanent discontinuation of study product because of safety or tolerability reasons.

Exclusion Criteria (Part A and B):

* Severe or unstable systemic sclerosis
* Significant diseases or conditions other than systemic sclerosis that may influence response to the study product or safety;
* Any one of the following values for laboratory tests at Screening:

  1. A positive pregnancy test (or at Visit 1);
  2. Hemoglobin < 10 g/dL
  3. Neutrophils < 1.0 x 10^9/L
  4. Platelets < 75 x 10^9/L
  5. Creatinine clearance < 50 ml/min according to modified Cockcroft-Gault equation
  6. Serum transaminases > 2.0 x upper normal limit
  7. Total bilirubin ≥ 1.5 x upper limit of normal
* Any other condition that, in the opinion of the Principal Investigator, is clinically significant and may put the subject at greater safety risk, influence response to study product, or interfere with study assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiera, M.D., Principal Investigator — Weill Cornell Medical College, New York City, NY
Locations (9):
- United States (9):
  - Arthritis Association of Southern CA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - John Hopkins Scleroderma Center, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Rutgers University, New Brunswick, New Jersey
  - Weill Cornell Medical College, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Houston Medical School, Houston, Texas
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenabasum (JBT-101) 5 mg QD/20 mg BID: Lenabasum 5 mg QAM and placebo QPM on Days 1-28, then lenabasum 20 mg BID on Days 29-84.
- Lenabasum (JBT-101) 20 mg QD/20 mg BID: Lenabasum 20 mg QAM and placebo QPM on Days 1-28, then lenabasum 20 mg BID on Days 29-84.
- Lenabasum (JBT-101) 20 mg BID/20 mg BID: Lenabasum 20 mg BID on Days 1-84.
Period: Overall Study
Arm/Group | Lenabasum (JBT-101) 5 mg QD/20 mg BID | Lenabasum (JBT-101) 20 mg QD/20 mg BID | Lenabasum (JBT-101) 20 mg BID/20 mg BID | Placebo
Started | 9 | 9 | 9 | 15
Completed | 8 | 8 | 8 | 14
Not Completed | 1 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenabasum (JBT-101) 5 mg QD/20 mg BID | Lenabasum (JBT-101) 20 mg QD/20 mg BID | Lenabasum (JBT-101) 20 mg BID/20 mg BID | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 15 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 7 | 15 | 39
  >=65 years | 1 | 0 | 2 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (10.75) | 47.2 (4.63) | 49.1 (14.57) | 46.5 (11.05) | 47.9 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 6 | 9 | 32
  Male | 0 | 1 | 3 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 5
  Not Hispanic or Latino | 8 | 7 | 7 | 14 | 36
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 6 | 8 | 8 | 12 | 34
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 9 | 15 | 42
Baseline Modified Rodnan Skin Score (mRSS) [Mean (Standard Deviation); unit: units on a scale] — The mRSS is an evaluation of patient's skin thickness by clinical palpation using a 0-3 scale; 0 = normal skin; 1 = mild thickness; 2 = moderate thickness; 3 = severe thickness with inability to pinch the skin into a fold for each of 17 surface anatomic areas of the body: face, anterior chest, abdomen, and, with right and left sides of the body separately evaluated, the fingers, forearms, upper arms, thighs, lower legs, dorsum of hands and feet. Individual values are summed and defined as the total skin score. Lowest score of 0 and maximum of 51 with higher scores indicate worse symptomology.
  units on a scale | 21.6 (9.29) | 26.7 (12.03) | 22.3 (10.16) | 26.2 (11.12) | 24.5 (10.60)
Baseline HAQ-DI [Mean (Standard Deviation); unit: units on a scale] — Health Assessment Questionnaire - Disability Index includes 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are two or three questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). The eight scores of the eight sections are summed and divided by 8. If one section is not completed by a subject, the summed score is divided by 7. As such, maximum scores can vary with a min of 0. The result is the DI, the disability index or functional disability index. Higher scores indicate worse symptomology.
  units on a scale | 1.07 (0.745) | 1.49 (0.697) | 0.83 (0.890) | 1.51 (0.793) | 1.26 (0.809)
Baseline FVC % Predicted [Mean (Standard Deviation); unit: percent predicted] — Population: Note: One subject in the Placebo cohort did not have a FVC % predicted measurement conducted, as such, the total number of subjects in the placebo cohort for FVC % predicted is n = 14 and for the total population, n = 41.
  percent predicted
    number analyzed (Participants) | 9 | 9 | 9 | 14 | 41
    (all) | 84.15 (9.044) | 93.79 (11.740) | 80.10 (15.993) | 79.61 (10.286) | 84.33 (12.185)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events From Baseline at Day 113
Description: The overall number of subjects with TEAE's per treatment group during active dosing (Days 1-84) plus the 28 day follow-up.
Time Frame: Part A: Day 113
Population: Per the statistical analysis plan, the intent was to analyze all subjects receiving lenabasum and compare to those subjects receiving placebo for the primary endpoint. As such, individual lenabasum groups were not reported to follow the pre-specified statistical analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Combined Lenabasum Group: Combination of all lenabasum cohorts for analysis purposes only.
Arm/Group | Placebo | Combined Lenabasum Group
Number analyzed (Participants) | 15 | 27
Participants | 9 | 17

2. Primary Outcome: Combined Response Index in Diffuse Cutaneous Systemic Sclerosis (CRISS) at Day 85 and 113
Description: CRISS components included the following domains: modified Rodnan skin score, forced vital capacity percent predicted, Physician Global Assessment, Patient Global Assessment, and Health Assessment Questionnaire Disability-Index. An algorithm determines the predicted probability of improvement from baseline by incorporating change in the mRSS, FVC percent predicted, Physician and Patient Global Assessments, and HAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A cut-off at 0.6 in the predicted probability of being improved has yielded the smallest misclassification error. Subjects are not considered improved if, between Visit 1 and 6, they develop new: 1) renal crisis; 2) decline in FVC% predicted by 15% (relative) from baseline and confirmed after 1 month; or 3) left ventricular failure (systolic ejection fraction < 45%) or pulmonary artery hypertension. Higher CRISS scores indicates improvement.
Time Frame: Day 85 and Day 113
Population: Per the statistical analysis plan, the intent was to analyze all subjects receiving lenabasum and compare to those subjects receiving placebo for this endpoint. As such, individual lenabasum groups were not reported to follow the pre-specified statistical analysis plan. Only subjects with values at Visit 5 and 6 were included in this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | Combined Lenabasum Group
Number analyzed (Participants) | 15 | 26
units on a scale
  CRISS score at Visit 5 (Day 85) | 0.010 [0.00 to 1.00] | 0.275 [0.00 to 1.00]
  CRISS score at Visit 6 (Day 113) | 0.00 [0.00 to 1.00] | 0.330 [0.00 to 1.00]

3. Secondary Outcome: CRISS Individual Components (mRSS Total Score) Change From Baseline.
Description: The LS mean change from baseline (CFB) at Visit 5 (Day 85) and 6 (Day 113) is provided for mRSS total score. Change from Change from Baseline was calculated as Visit 5 - Baseline and independently Visit 6 - Baseline. The mRSS consists of an evaluation of patient's skin thickness rated by clinical palpation using a 0-3 scale (0 = normal skin; 1 = mild thickness; 2 = moderate thickness; 3 = severe thickness with inability to pinch the skin into a fold for each of 17 surface anatomic areas of the body: face, anterior chest, abdomen, and, with right and left sides of the body separately evaluated, the fingers, forearms, upper arms, thighs, lower legs, dorsum of hands and feet. Individual values are summed and defined as the total skin score. Total score is 0 to 51 with higher scores indicating worse symptomology
Time Frame: Day 85 and 113
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Combined Lenabasum Cohorts: This analysis group combines data from lenabasum Cohort 1 (5 mg QD/20mg BID), Cohort 2 (20 mg QD/20 mg BID), and Cohort 3 (20 mg BID/20 mg BID) for analysis purposes only.
- Placebo: Placebo subjects in this study received placebo for the entire duration of the trial.
Arm/Group | Combined Lenabasum Cohorts | Placebo
Number analyzed (Participants) | 27 | 15
units on a scale
  mRSS Total Score CFB at Visit 5 (Day 85) | -3.8 (1.1) | -2.6 (1.5)
  mRSS Total Score CFB at Visit 6 (Day 113) | -4.7 (1.1) | -2.0 (1.5)

4. Secondary Outcome: CRISS Individual Component (FVC Percent Predicted) Change From Baseline
Description: The LS mean change from baseline (CFB) at Visit 5 (Day 85) and 6 (Day 113) is provided for FVC percent predicted. Change from Baseline was calculated as Visit 5 - Baseline and independently Visit 6 - Baseline.
Time Frame: Day 85 and 113
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Combined Lenabasum Cohorts | Placebo
Number analyzed (Participants) | 27 | 15
percent predicted
  FVC % predicted CFB at Visit 5 (Day 85) | 0.90 (0.99) | -0.77 (1.32)
  FVC % predicted CFB at Visit 6 (Day 113) | 0.20 (0.92) | -0.98 (1.22)

5. Secondary Outcome: CRISS Individual Component (Physician Global Assessment Score) Change From Baseline
Description: The LS mean change from baseline (CFB) at Visit 5 (Day 85) and 6 (Day 113) is provided for physician global assessment. Change from Baseline was calculated as Visit 5 - Baseline and independently Visit 6 - Baseline. The Physician Global Assessment of disease activity will be performed using a segmented numerical version of the visual analogue scale in which the physician selects a whole number (0-10 integers) that best reflects the overall disease activity. The numerical rating score is anchored by 2 verbal descriptors, one of "no disease activity" (score of 0) and one of "worse imaginable disease activity" (score of 10), with numbers 1-9 spaced equidistance in between. The physician will select an integer to describe disease activity. The recall period is one week.
Time Frame: Day 85 and 113
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Lenabasum Cohorts | Placebo
Number analyzed (Participants) | 27 | 15
units on a scale
  Physician Global Assessment Score CFB at Visit 5 | -0.9 (0.3) | -0.5 (0.4)
  Physician Global Assessment Score CFB at Visit 6 | -0.9 (0.3) | -0.7 (0.3)

6. Secondary Outcome: CRISS Individual Component (Patient Global Assessment Score) Change From Baseline
Description: The LS mean change from baseline (CFB) at Visit 5 (Day 85) and 6 (Day 113) is provided for patient global assessment. Change from Baseline was calculated as Visit 5 - Baseline and independently Visit 6 - Baseline. The assessment at each specified visit will be performed with a segmented numerical version of the visual analogue scale in which the subject selects a whole number (0-10 integers) that best reflects the overall disease activity. The numerical rating score is anchored by two verbal descriptors, one of "no disease activity" (score of 0) and one of "worse imaginable disease activity" (score of 10), with numbers 1-9 spaced equidistance in between. The subject will select an integer to describe disease activity. The recall period is one week.
Time Frame: Day 85 and 113
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Lenabasum Cohorts | Placebo
Number analyzed (Participants) | 27 | 15
units on a scale
  Patient Global Assessment Score CFB at Visit 5 | -0.8 (0.4) | 0.4 (0.6)
  Patient Global Assessment Score CFB at Visit 6 | -0.9 (0.4) | 0.3 (0.5)

7. Secondary Outcome: CRISS Individual Component (HAQ-DI Score) Change From Baseline.
Description: Change from Baseline was calculated as Visit 5 - Baseline and independently Visit 6 - Baseline. Health Assessment Questionnaire - Disability Index includes 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are two or three questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). The eight scores of the eight sections are summed and divided by 8. If one section is not completed by a subject, the summed score is divided by 7. As such, maximum scores can vary with a min of 0. The result is the DI, the disability index or functional disability index. Higher scores indicate worse symptomology
Time Frame: Day 85 and 113
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Lenabasum Cohorts | Placebo
Number analyzed (Participants) | 27 | 15
units on a scale
  HAQ-DI CFB at Visit 5 (Day 85) | -0.22 (0.07) | 0.11 (0.10)
  HAQ-DI CFB at Visit 6 (Day 113) | -0.14 (0.07) | 0.11 (0.09)

ADVERSE EVENTS:
Time Frame: Days 1 - 113
Description: Lenabasum (JBT-101) 5 mg QD/20 mg BID, Lenabasum (JBT-101) 20 mg QD/20 mg BID, and Lenabasum (JBT-101) 20 mg BID/20 mg BID Groups were combined (i.e., Combined Lenabasum) as pre-specified in the study protocol.
Groups:
- Placebo (Days 1 - 84 + After-treatment Period): Placebo cohort for the overall study.
- Combined Lenabasum (Days 1 - 84 + After-treatment Period): Combined lenabasum cohorts for the overall study.
Arm/Group | Placebo (Days 1 - 84 + After-treatment Period) | Combined Lenabasum (Days 1 - 84 + After-treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/27
Other Adverse Events (participants affected / at risk) | 9/15 | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Days 1 - 84 + After-treatment Period) (N=15) | Combined Lenabasum (Days 1 - 84 + After-treatment Period) (N=27)
Vomiting (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Days 1 - 84 + After-treatment Period) (N=15) | Combined Lenabasum (Days 1 - 84 + After-treatment Period) (N=27)
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1 — and administration site conditions
Fatigue (General disorders) | 1 | 5
Feeling abnormal (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Small intestinal bacterial overgrowth (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Forced vital capacity decreased (Investigations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 6
Headache (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Uticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischemia (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes